CLINICAL TRIAL: NCT04174326
Title: Cognitive Behavioral Pain Management Program for Children and Youth With Cerebral Palsy (CBPM_CP): a Feasibility Study
Brief Title: CBT Program for Pain Management for Children and Youth With CP (CBT=Cognitive Behavioral Therapy; CP= Cerebral Palsy)
Acronym: CBT;CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB19-850
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy; Chronic Pain
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Cerebral Palsy; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either immediate treatment group or delayed waitlist treatment group at baseline. Participants in both groups will receive the same CBT intervention program consecutively, once a week during a period of 6 weeks. Two in-between sessions practice assignments will be included in each therapy session in the program. Participants will be followed-up at 18 weeks from the beginning of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A weekly 2 hour CBT for chronic pain group intervention for a duration of 6 weeks
  Interventions: Behavioral: Immediate intervention group
- Delayed intervention group (No Intervention): A waiting list for CBT for chronic pain group intervention.

INTERVENTIONS:
Behavioral: Immediate intervention group — Participants will be randomized to either the immediate or delayed intervention group at baseline. Participants in both groups will receive CBT for chronic pain management sequentially, once a week during the 6 week intervention period. Participants will be followed-up at 18 weeks from baseline. Two in-between sessions practice assignments will be added to each group therapy session during the the CBT program.
  Other Names: Immediate
  Arms: Intervention group

SUMMARY:
This study will focus on the feasibility of a modified cognitive behavioral program for pain management among children and youth with cerebral palsy (CP) on developing pain coping skills and reducing pain interference levels The study design is a randomized control feasibility trial. Participants will be placed randomly into one of two groups based on chance (50/50). The 2 groups are: (1) immediate treatment group and (2) delayed wait-list treatment group.

Both groups will receive the same intervention protocol.

DETAILED DESCRIPTION:
Children with CP often experience pain that is related to their medical condition and that may limit or interfere with their everyday activities and Quality of Life (QoL).One possible way to help these children is by using a modified cognitive behavioral therapy (CBT) for pain management.

For this study, the investigators want to do a feasibility study, to see if participating in a six-week pain management CBT program for children and youth with CP and their parents, leads to better pain coping skills and lower levels of pain interference, when compared to a controlled waiting list.

Participants in both groups (immediate and delayed treatment) will participate in a 2-hour CBT session, once a week, for a total of six weeks. Following 3-months from the last CBT session, participants will be contacted for a short follow-up screening. All participants will be enrolled in the study for a total of 18 weeks.

This study will be done at the Holland Bloorview Kids Rehabilitation Hospital, Toronto, Canada. Sixteen participants with CP (gross motor function classification system (GMFCS) levels I-V), age 8 to 18, with evidence of chronic pain (detailed as pain lasting more than 3 months or lasting longer than the expected time to heal) and their parents, will be recruited for participation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CP
2. Chronic pain lasting greater than 3 months and restricting some or all activities according to child/youth/parental self-report
3. A baseline score of 70 (~ -2 SD) on each of the three vineland adaptive behavior scales (VABS) sub-scales: communication, daily living skills and socialization
4. Successful completion of a modified sorting task including sorting cubes according to size and rating activities in order of how much they like to do them
5. Parent agreement to participate in the parents' program
6. Can communicate in English, with or without the use of augmentative communication devices

Exclusion Criteria:

Participants who meet any of the following criteria will not be eligible to take part in the trial:

1. Diagnosis of major visual or hearing impairment
2. Currently attending psychological treatment focused on pain management; (3) Uncontrolled seizure(s) (with or without medication) in the previous 12 months.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pediatric Pain Interference Scale [PPIS] | Changes in PPIS from baseline to 6 and 18 weeks
  The Pediatric Pain Interference Scale (PPIS) was developed by the National Institutes of Health Patient Reported Outcomes Measurement Information System (PROMIS) initiative. The scale assesses pain-related behaviors across 5 domains (pain, fatigue, physical functioning, social health, and emotional health) and has been validated with pediatric populations (5-18 years) representing a variety of chronic health conditions, including CP. Scores vary from 8 to 40 with higher scores indicating higher level of pain interference. Decrease in levels of pain interference is considered a better outcome.
Proportion of eligible participants that are recruited as study participants during the study timeline [Feasibility] | 18 weeks
  Participants must meet all eligibility criteria in order to be included in the analysis of this outcome measure. A higher proportion of eligible patients recruited is considered to be a better outcome.
Proportion of recruited participants that attend in 80% of the 6 study sessions during the intervention phase [Feasibility] | 18 weeks
  Number of sessions participants engage in during the intervention phase vs. total number of sessions in the program. Participants must attend at least 5 of 6 sessions to reach 80% adherence to CBT sessions. Higher participation rate in therapy is considered to be a better outcome.
Proportion of recruited participants that completed 80% of the in-between session assignments during the intervention phase [Feasibility]. | 18 weeks
  Adherence to in-between sessions assignments score will be calculated based on number of assignments completed vs. anticipated compliance during the intervention phase (a total of 12 assignments). Higher adherence to complete in-between session assignments during therapy is considered to be a better outcome.
Proportion of recruited participants that attended the follow-up session 18 weeks from baseline [Feasibility]. | 18 weeks
  Adherence to participate in the follow-up session following the completion of the treatment. Higher adherence to participate in follow-up sessions is considered to be a better outcome.

SECONDARY OUTCOMES:
The Faces Pain Scale-Revised [FPS-R] | Changes in pain intensity from baseline to 6 and 18 weeks
  The Faces Pain Scale - Revised [FPS-R] is a self-report measure of pain intensity developed for children. The scale shows a close linear relationship with visual analog pain scales across the age range of 4-16 years. It is easy to administer and requires no equipment except for the photocopied faces. Numerical self-rating scales (0-10, with "0" equals "No pain" and "10" equals "Very much pain") can be used with most children older than 8 years of age and behavioral observation scales are required for those unable to provide a self-report. Decrease in pain intensity is considered a better outcome
Psychological Inflexibility in Pain Scale [PIPS] | Changes in pain coping from baseline to 6 and 18 weeks
  The Psychological Inflexibility in Pain Scale (PIPS) is a screening tool used to measure pain willingness and activities engagement of individuals living with chronic pain. It emphasizes the willingness to experience pain rather than trying to control or reduce pain symptoms. The tool was developed for adults and has been used with children and adults ages 8 - 84 years. It is a 16- item tool that consists of two subscales, avoidance and cognitive function. Participants rate how true the statements are on a 7-point Likert scale ranging from 'never true' to 'always true', with mean scores ranging from 1-7. Higher scores indicate greater levels of psychological inflexibility. Decrease in pain inflexibility is considered a better outcome
KIDSCREEN-27 Health related quality of life [HRQoL] | Changes in HRQoL from baseline to 18 weeks
  The KIDSCREEN-27 questionnaire will be used for evaluating Health related quality of life. The questionnaire consists of 27 items which are used to assess HRQoL across 5 dimensions: Physical Well-Being (5 items); ; Psychological Well-Being (7 items) ; Parent Relations & Autonomy (7 items); Social Support & Peers (4 items), and; School Environment (4 items). The items assess either the frequency of behavior/feelings or, in fewer cases, the intensity of an attitude and are answered on a five-point scale. Mean scores range between 1-5 with higher values indicating higher health related quality of life. Increase in health related quality of life is considered a better outcome.
Pain Stages of Change Questionnaire-Parents [PSOCQ-P] | Changes in PSOCQ-P from baseline to 18 6 and weeks
  Pain Stages of Change Questionnaire will be used to assess parents' own levels of readiness to encourage their child to adopt a self-management approach to pain treatment. The Pain Stages of Change Questionnaire-Parents (PSOCQ-P) yields four validated subscales: Precontemplation, Contemplation, Action, and Maintenance, with precontemplation being the least ideal and indicating no consideration by the parent of having the child adopt a self-management approach to pain treatment. Mean scores on each scale range between 1 to 5, with higher scores indicating stronger endorsement of items representing each readiness stage domain. A decrease in Precontemplation and Contemplation scores and increase in Action and Maintenance scores indicate better outcome.
Chronic Pain Acceptance Questionnaire-Parent [CPAQ-P] | Changes in CPAQ-P from baseline to 6 and 18 weeks
  The Chronic Pain Acceptance Questionnaire- (parent version) (CPAQ-P) assesses parents' beliefs about child's acceptance of pain. The CPAQ-P consists of 16 items scored on a Likert scale of 0 = "never true" to 6 = "always true". The 16 items comprise two subscales: Activity Engagement (9 items) and Pain Willingness (7 items). Activity engagement reflects the degree of participation in regular daily activities in the presence of pain (e.g. "My life is going well, even though I have chronic pain"). Pain willingness reflects the absence of attempts to avoid or control pain (e.g. "I avoid putting myself in situations where my pain might increase" - reverse keyed). Mean scores on each scale range between 1-6. Higher scores on both scales indicate greater parental beliefs about child acceptance of pain. An increase in scores on both scales is considered a better outcome.

OTHER OUTCOMES:
Canadian Occupational Performance Measure [COPM] | Changes in COPM from baseline to 18 weeks
  Achievement of individualized goals will be evaluated using the [COPM]. Each participant will set a COPM individualized goal related to an aspect of activity that has pain interference (e.g. improved sleep, improved seating tolerance). The client is asked to use a 10 point scale to rate their own level of performance and satisfaction with performance for each of the identified problems. The therapist calculates an average COPM performance score and satisfaction score. These typically range between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction. Research evidence suggests that a change of two or more points on performance and satisfaction scales represents a clinically important change.
Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider [PRIME-SP] | Change in engagement in intervention session from baseline to 18 weeks.
  Service provider observations (i.e., psychologist/ social worker) of participants' engagement in the intervention sessions, will be evaluated using the Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider (PRIME-SP). Engagement scores range between 1= "disengaged" to 4= "extremely engaged", with higher mean scores indicating higher engagement. In addition, service providers rate clients affective, behavioral and cognitive involvement in sessions, ranging from 1= "not at all" to 4= "to a great extent". Higher scores indicate higher involvement in each domain.
  Increase in participant's engagement and involvement is considered a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Fehlings, MD, MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland-Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No